CLINICAL TRIAL: NCT06672822
Title: An Open Label Evaluation of Intralesional Injection of Sodium Thiosulfate in the Treatment of Cutaneous or Tendon Calcinosis in Connective Tissue Disease
Brief Title: Intralesional Injection of STS in Treatment of Calcinosis
Acronym: STSINJ
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Robyn T. Domsic, MD, MPH (Other)
Collaborators: National Institute of Arthritis and Musculoskeletal and Skin Diseases (NIAMS) (NIH)
Responsible Party: Sponsor-Investigator, Robyn T. Domsic, MD, MPH, Associate Professor, University of Pittsburgh
Organization: University of Pittsburgh (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: STUDY24040146; 5P50AR080612 (NIH)
Record Dates: First submitted 2024-10-30; First posted 2024-11-04 (Actual); Last update posted 2025-09-08 (Actual); Status verified 2025-03

CONDITIONS: Systemic Sclerosis (SSc); Dermatomyositis; Mixed Connective Tissue Disease (MCTD); Calcinosis
Keywords: calcinosis
MeSH Terms: conditions — Scleroderma, Systemic; Dermatomyositis; Mixed Connective Tissue Disease; Calcinosis | interventions — sodium thiosulfate

STUDY DESIGN:
Intervention Model Description: Open label, single-arm, single center US study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Sodium thiosulfate (STS) (Experimental): Open label, single-arm, receiving 1-5ml of STS (250mg/ml) sodium thiosulfate (STS) injections to calcinosis lesions.
  Interventions: Drug: Sodium Thiosulfate (STS)

INTERVENTIONS:
Drug: Sodium Thiosulfate (STS) — Depending on the size of the calcinosis lesion, 1-5ml of STS (250mg/ml) will be used for injection under ultrasound guidance.

SUMMARY:
The specific objective of this study is to perform a small, open-label study to assess the safety and efficacy of intralesional, subcutaneous injection of STS on calcinosis symptoms and lesion size in systemic sclerosis (SSc), mixed connective tissue disease (MCTD) and dermatomyositis (DM) patients. Injection will be guided by ultrasound, lesion size assessed by ultrasound, and symptom burden by patient-reported outcome measures.

DETAILED DESCRIPTION:
Calcinosis is a condition in which calcium builds up in the skin and tissue under the skin. It develops in ∼30% of adult dermatomyositis,18%-49% of systemic sclerosis patients, 25-40% of patients with limited systemic sclerosis. There is no standard treatment recommended by physicians currently. Many treatments have been tested, all with limited benefits and without good evidence that any are effective. They are, based only on single cases or small numbers of patients in studies called "case series." But in some cases, these agents may be effective.

There are several case series that have shown the effectiveness of injecting a chemical compound called sodium thiosulfate (or "STS") into calcinosis lesions. There was some improvement in terms of pain control, and a decrease in size and resolution of the calcinosis. The aim of our study is to test intralesional sodium thiosulfate (STS) injection for symptoms relief of calcinosis. STS has been approved by the U.S. Food and Drug Administration for certain conditions related to childhood cancers. It has not been approved by the FDA to treat calcinosis. The specific aims of this study are to assess change in calcinosis size and quality-of-life measures.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of systemic sclerosis, mixed connective tissue disease or inﬂammatory myopathy
* Must be over 18 years of age
* Participants must be competent to give informed consent
* Participants must have radiographic evidence (xray or ultrasound) of calcinosis.
* Participants must need symptomatic relief

Exclusion Criteria:

• Pregnant women will be excluded

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2025-03-17 (Actual); Primary Completion 2028-08-31 (Estimated); Study Completion 2029-05-01 (Estimated)

PRIMARY OUTCOMES:
Primary endpoint: Change in size of calcinosis lesion from baseline to 12 weeks | 12 weeks
  Change in size of calcinosis lesions will be measured by x-ray at baseline and then again at 12 weeks.

SECONDARY OUTCOMES:
Change in pain (interference) | up to 12 weeks
  We will evaluate pain impact on quality-of-life using the PROMIS® (Patient-Reported Outcomes Measurement Information System) Pain Interference Short Form 4a. This is a 4-question patient-reported outcome measure asking patients about their experience in the last week. Responses are in a likert scale format from 'not at all' to 'very much' Higher scores indicate higher degrees of interference with important aspects of life. The raw score is converted to a T-score with a mean of 50 and a standard deviation (SD) of 10.
Change in Pain Intensity | up to 12 weeks
  We will measure pain intensity using the PROMIS® Pain Intensity 3a scale. This is a 30-item questionnaire inquiring about pain over the last week. Higher scores indicate higher pain intensity. Raw scores are converted to a T-score for analysis. The t-score is set to a mean of 50 and a standard deviation (SD) of 10.
Health-related Quality of Life using the EQ-5D-5L | up to 12 weeks
  EuroQol(EQ)-5D-5L is a validated self-reported patient questionnaire assessing five domains of health quality: pain/discomfort, mobility, self-care, activity and anxiety/depression plus a patient global assessment visual analog scale (VAS). Patients can report no, some problems or extreme problems (scored 1-3); the VAS is scored 0-100. Iull health is a score of 1 and values below zero are regarded as a state worse than death.
Scleroderma Health Assessment Questionnaire (SHAQ) | up to 12 weeks
  The SHAQ is composed of the standard Health Assessment Questionnaire (HAQ-DI)) plus additional visual analog scales to measure symptoms important in scleroderma: vascular, digital ulcers, lung, gastrointestinal, pain and patient global assessment. The HAQ-DI questions are scored 0-3. Higher scores indicate greater disability.
Change in calcinosis related symptom severity | up to 12 weeks
  The Mawdsley calcinosis scale consists of Part A and Part B. Part A asks about presence of calcinosis or ulcers overlying calcinosis. If the response is present, then Part B is completed. Part B consists of 17 questions inquiring over the last 2 weeks of symptoms. Responses are 0-10 from no limitation/not all to maximum/worst possible. Higher scores indicate higher symptom severity from calcinosis.

CONTACTS AND LOCATIONS:
Overall Officials: Robyn T Domsis, MD, Principal Investigator — University of Pittsburgh
Locations (1):
- UPMC Arthritis and Autoimmunity Center, Pittsburgh, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: Yes
Data should be requested by contacting the P0I once results are published. Data sharing will conform to all local and federal regulations and be de-identified with data use agreements in place.

REFERENCES:
- [Background] Boulman N, Slobodin G, Rozenbaum M, Rosner I. Calcinosis in rheumatic diseases. Semin Arthritis Rheum. 2005 Jun;34(6):805-12. doi: 10.1016/j.semarthrit.2005.01.016. PMID 15942915
- [Background] Chander S, Gordon P. Soft tissue and subcutaneous calcification in connective tissue diseases. Curr Opin Rheumatol. 2012 Mar;24(2):158-64. doi: 10.1097/BOR.0b013e32834ff5cd. PMID 22227955